CLINICAL TRIAL: NCT05323864
Title: Going to Altitude With Anxious-depressive Symptoms - a Randomised Cross Over Trial in Individuals With Mental Disorders and Healthy Controls
Brief Title: Going to Altitude With Anxious-depressive Symptoms
Acronym: Psychoxie
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022
Record Dates: First submitted 2022-02-21; First posted 2022-04-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hypoxia; Mental Disorder
Keywords: anxiety; depressive symptoms; high altitude
MeSH Terms: conditions — Hypoxia; Mental Disorders; Anxiety Disorders; Depression; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled crossover trial with two groups of participants will be conducted. One group will be a group of psychiatric patients and the other group will be a group of healthy controls. The study will follow a crossover design with random allocation of condition order (i.e., normobaric hypoxia or sham hypoxia).
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric hypoxia (Experimental): Normobaric hypoxia equivalent to 3800m terrestrial altitude. The chamber located on the campus of the University of Innsbruck's Department of Sport Science. The chamber dimension is 5 x 3m.
  Interventions: Biological: Hypoxia
- Sham hypoxia (Sham Comparator): The chamber located on the campus of the University of Innsbruck's Department of Sport Science. The chamber dimension is 5 x 3m.
  Interventions: Biological: Hypoxia

INTERVENTIONS:
Biological: Hypoxia — Participants will be randomly assigned to start with the normobaric hypoxia condition or the sham hypoxia condition. They will swap to the other condition during the second visit, which will be executed at least 14 days after the first visit. Each sojourn will last for six hours and participants will reside in the chamber individually. During the six-hour stay, participants will be allowed to move freely within the chamber.

SUMMARY:
Introduction: Currently, there is a lack of international guidelines or clinical recommendations for individuals with mental illnesses (i.e., bipolar disorder, posttraumatic stress disorder) going on high altitude sojourns. However, these guidelines would be important considering that mental illnesses are among the most common disorders worldwide and millions of people are hiking at high altitudes in the Alps, being granted easy access up to 3800m by cable cars. Before conceptualizing these guidelines, it seems necessary to study the physiological and psychological effects of ambient pressure changes leading to oxygen deficiency (hypoxia) in individuals with mental illnesses when being exposed to hypoxic conditions. The investigators hypothesize a shift towards negative affective responses and state anxiety as well as increased levels of neurotransmitter precursor amino acids (PHE/TYR and KYN/TRP) in individuals with mental illnesses when being exposed to hypoxic conditions.

Methods and Analysis: The investigators plan to perform a double-blind randomized controlled trial in a safe laboratory environment by using a normobaric hypoxic chamber. Participants suffering from depression and anxiety symptoms will be included as well as age and sex-matched healthy controls. They will attend a six-hour exposure equivalent to 3800m of altitude as well as a six-hour exposure to sham hypoxic conditions. Recruited participants will be screened by the Beck Anxiety and Depression Inventory, the Symptom Checklist (SCL-90) as well as an interview assessment. Affective responses in state anxiety will be assessed before, and during each hour of exposure by using the Feeling Scale (FS), Felt Arousal Scale (FAS), Positive and Negative Affect Schedule (PANAS), State-Anxiety Inventory (STAI) and subjective mental stress levels (Visual Analogue Scale; VAS). Physiological parameters will be assessed by venous blood sampling, pulse oximetry and oxidative stress level measurement before entering the chamber, after three and six hours of exposure. Additionally, symptoms of acute mountain sickness will be assessed by the Lake Louise Score before, after three and six hours of exposure. Follow-up measurements are planned one and seven days after the chamber visit, consisting of venous blood sampling, the Beck Anxiety and Depression Inventory.

A series of univariate analyses of covariance (ANCOVA) for repeated measures will be used to test the three-way (i.e. "group × condition × time") and two-way ("group × condition" and "group × time") interactions. Analyses will be adjusted for possible confounding, by adding age, sex, smoking, prior AMS, and medication status in the models as covariates.

Ethics and dissemination: Ethical approval has been obtained from the ethics committee of the Medical University of Innsbruck (1250/2021).

ELIGIBILITY:
Inclusion Criteria:

* sufficient command of the German language
* no psychotic or cognitive disorders
* patients suffering from anxious-depressive symptoms (meeting the cut off points of light-medium in the screening for anxiety and depression symptoms)

Exclusion Criteria:

* pregnant or breastfeeding
* permanent residence above 1000m
* overnight stays at altitudes above 2500m in the previous month
* exposure to 2500m or higher two weeks prior to the six-hour hypoxic exposure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in affective responses | up to 6 hours, including 8 measurements, measuring before the start of intervention, every hour during the intervention, and after the end of intervention
  Self-reported questionnaire to assess affective valence, perceived activation, positive and negative affect
Changes in state anxiety | up to 6 hours, including 8 measurements, measuring before the start of intervention, every hour during the intervention, and after the end of intervention
  Self-reported questionnaires to assess state anxiety
Changes in subjective perception of stress | up to 6 hours, including 8 measurements, measuring before the start of intervention, every hour during the intervention, and after the end of intervention
  Self-reported questionnaires to assess subjective perception of stress

SECONDARY OUTCOMES:
Changes in anxious-depressive symptoms | 10 days, including 3 measurements at baseline, day 1 and follow-up day 7
  Self-reported questionnaires to assess depression symptoms, anxiety symptoms, and subjectively perceived impairment due to physical and psychological symptoms
Changes in inflammatory parameters CRP | 8 days, including 4 measurements pre intervention, after 3 hours of intervention, at the end of intervention (6 hours), and at follow-up after 7 days
  Venous blood samples to assess CRP (C-reactive protein)
Changes in inflammatory parameters IL-6 | 8 days, including 4 measurements pre intervention, after 3 hours of intervention, at the end of intervention (6 hours), and at follow-up after 7 days
  Venous blood samples to assess IL-6 (interleukin 6)
Changes in oxidative stress | 6 hours, including 3 measurements, measuring pre intervention, after 3 hours of intervention, at the end of intervention (6 hours)
  Capillary blood samples from the fingertip collected with the Free Carpe Diem device by DIACRON International to measure total antioxidant capacity and the antioxidant potential of plasma

CONTACTS AND LOCATIONS:
Locations (1):
- University of Innsbruck, Department of Sport Science, Innsbruck, Tyrol, Austria